CLINICAL TRIAL: NCT05861453
Title: An Open-label Mechanistic Study to Assess the Pharmacokinetics, Pharmacodynamics and Safety of Orally Administered Epeleuton in Patients With Sickle Cell Disease
Brief Title: Pharmacokinetics, Pharmacodynamics and Safety of Epeleuton in Patients With Sickle Cell Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Afimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS102A-10-RD2
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — epeleuton

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epeleuton 4g/day (Experimental)
  Interventions: Drug: Epeleuton

INTERVENTIONS:
Drug: Epeleuton — Participants will receive 2000mg Epeleuton (DS102) capsules twice daily.
  Other Names: DS102 Capsules

SUMMARY:
To assess the pharmacokinetics, pharmacodynamics and safety of Epeleuton capsules in adult SCD patients who are aged ≥18 years.

DETAILED DESCRIPTION:
The trial will consist of a 28-day screening period, 16 weeks of active treatment and a 30-day post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease (SCD) including:

  * 2 sickle hemoglobin genes [HbSS]
  * HbSβ0 thalassemia
  * HbSβ+ thalassemia
  * Heterozygous for hemoglobin S and hemoglobin C [HbSC]
* Male or female patients aged 18 years and older on the day of signing the informed consent form (ICF)
* Patients who have had between 2 and 15 episodes of vaso-occlusive crisis (VOC) in the past year (12 months)
* For patients taking hydroxyurea (HU), the dose of HU must be stable for at least 3 months prior to signing the ICD and with no anticipated need for dose adjustment during the study.
* Female patients and male patients with female partners of childbearing potential must use highly effective contraceptive methods for the duration of the study.

Exclusion Criteria:

* Patients who are receiving regularly scheduled blood (RBC) transfusion therapy (also termed chronic, prophylactic, or preventive transfusion), have received an RBC transfusion for any reason within three months of the baseline visit
* Patients who have received a hematopoietic stem cell transplant.
* Patients with inadequate venous access as determined by the Investigator
* Patients who are pregnant, planning pregnancy, breastfeeding and/or are unwilling to use adequate contraception during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in P-selectin | 16 Weeks
  Change in P-selectin from baseline at Week 16.
Changes from baseline in Hemoglobin | 16 Weeks
  Change in hemoglobin from baseline at Week 16
Changes from baseline in absolute reticulocyte count | 16 Weeks
  Change in absolute reticulocyte count from baseline at Week 16.
Changes from baseline in E-selectin | 16 Weeks
  Change in E-selectin from baseline at Week 16.
Changes from baseline in Phosphatidylserine | 16 Weeks
  Change in Phosphatidlyserine from baseline to week 16.
Changes from baseline in annualized rate of VOCs leading to a healthcare visit, and VOCs that are treated at home | 16 Weeks
  Changes in annualized rate of VOCs leading to a healthcare visit, and VOCs that are treated at home from baseline to week 16
Changes from baseline in RBC Laminin Adhesion | 16 Weeks
  Changes in RBC Laminin Adhesion from baseline to week 16
Changes from baseline in Leukocytes | 16 Weeks
  Changes in Leukocytes from baseline to Week 16
Changes from baseline in Vascular Cell Adhesion Molecule 1 (VCAM-1) | 16 Weeks
  Changes in VCAM-1 from baseline to Week 16
Changes from baseline in Dense Red Blood Cells | 16 Weeks
  Changes in Dense Red Blood Cells from baseline to Week 16
Changes from baseline in Osmoscan | 16 Weeks
  Changes in Osmoscan from baseline to Week 16
Changes from baseline in Oxygen Point of Sickling | 16 Weeks
  Changes in Oxygen Point of Sickling from baseline to Week 16
Changes from baseline in D-dimer | 16 Weeks
  Changes in D-dimer from baseline to Week 16
Change from baseline in PROMIS Pain Interference Short Form | 16 Weeks
  Change in PROMIS Pain Interference from baseline to Week 16
Change from baseline in PROMIS Physical Activity Short Form | 16 Weeks
  Change in PROMIS Physical Activity from baseline to Week 16
Trough plasma concentrations of total and unesterified 15 HEPE | 16 Weeks
  Trough plasma concentrations of total and unesterified 15 HEPE at baseline and Week 16
Determination of exploratory biomarkers from baseline | 16 Weeks
  Determination of exploratory biomarkers at baseline and Week 16

CONTACTS AND LOCATIONS:
Locations (18):
- United States (16):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - New England Sickle Cell Institute, UConn Health, Farmington, Connecticut
  - Medstar Health, Washington D.C., District of Columbia
  - Aflac Cancer and Blood Disorders Center, Children's Healthcare of Atlanta at Hughes Spalding, Atlanta, Georgia
  - Emory University - Georgia Comprehensive Sickle Cell Center, Atlanta, Georgia
  - Aflac Cancer and Blood Disorders Center, Children's Healthcare of Atlanta at Arthur M. Blank Hospital, Atlanta, Georgia
  - UI Health Sickle Cell Center, Chicago, Illinois
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - The Center for Cancer and Blood Disorders, A Division of American Oncology Partners, PA, Bethesda, Maryland
  - Kaiser Permanente Mid-Atlantic States, Largo, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Robert Wood Johnson Medical School Rutgers, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Jacobi Medical Center, The Bronx, New York
  - UNC Health, Chapel Hill, North Carolina
  - Science 37, Morrisville, North Carolina
- Canada (2):
  - St Paul's Hospital Hematology/Oncology Research, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No